CLINICAL TRIAL: NCT05795140
Title: A Multi-center, Single Arm, Open-label Extension Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Iptacopan in Participants With Atypical Hemolytic Uremic Syndrome (aHUS) Who Have Completed a Preceding Iptacopan Phase 3 Study in aHUS
Brief Title: Evaluate Long-term Safety, Tolerability and Efficacy of Iptacopan in Study Participants With aHUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023F12001B
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: aHUS; iptacopan; atypical hemolytic uremic syndrome; thrombotic microangiopathy; TMA; dialysis; CKD; eGFR; PE/PI; Complement 3 Glomerulopathy (C3G); IgAN; PNH
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Thrombotic Microangiopathies; Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iptacopan 200 mg (Experimental): Open label , single arm
  Interventions: Drug: Iptcaopan 200 mg

INTERVENTIONS:
Drug: Iptcaopan 200 mg — Open label, participant specific kits, hard gelatin capsules to be taken twice a day
  Other Names: LNP023

SUMMARY:
This is a multicenter, single arm, open-label, extension study to evaluate the long-term safety, tolerability, and efficacy of iptacopan in participants with aHUS.

DETAILED DESCRIPTION:
The extension study Baseline/Day 1 visit is equivalent to the End of Treatment visit of the parent study. The study will begin on Day 1 followed by on-site visits every 4 months during the study treatment period. A Safety Follow Up tele-visit must be conducted 7 days after last study treatment to collect information on Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the open label extension study
2. Willing and able to comply with the study Schedule of Activities
3. Participants who have completed the full study treatment period of any prior "Novartis sponsored" iptacopan Phase 3 clinical trial in aHUS, are still on iptacopan study treatment and derive benefit from it as per Investigator's judgement
4. Prior vaccinations against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections should be up to date (i.e., any boosters required should be administered according to local guidelines)

Exclusion Criteria:

1. Concomitant treatment with any complement inhibitor as well as concomitant treatment with any of the prohibited drugs
2. Any comorbidity or medical condition (including but not limited to any active systemic bacterial, viral or fungal infection or malignancy) that, in the opinion of the Investigator could put the participant at risk
3. Active infection or history of recurrent invasive infections caused by encapsulated bacteria such as Neisseria meningitidis, Streptococcus pneumoniae or Haemophilus influenzae
4. History of hypersensitivity to iptacopan or its excipients or to drugs of similar chemical classes
5. Pregnant or nursing (lactating) women
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of investigational drug and for 1 week after stopping of investigational drug.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2032-12-23 (Estimated); Study Completion 2033-01-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Throughout the study duration, up to 4 years
  Number of participants with adverse events and serious adverse events will be provided
Number of participants with abnormal safety laboratory parameters, vital signs and ECGs | Throughout the study duration, up to 4 years
  Number of participants with abnormal safety laboratory parameters , vital signs and ECGs will be provided

SECONDARY OUTCOMES:
Number of participants with absence of aHUS relapse without the use of anti-C5 antibody | Throughout the study duration, up to 4 years
  Atypical hemolytic uremic syndrome (aHUS) relapse is defined by the coexistence of at least two of the following at the same visit:
  * thrombocytopenia (platelet count < 150 x 109 /L),
  * microangiopathic hemolytic anemia (hemoglobin < 10 g/dl, LDH > upper limit of normal, undetectable haptoglobin, presence of schistocyte on blood smear),
  * worsening kidney function (serum creatinine or urine protein to creatinine ratio (UPCR) > upper limit of normal and an increase of ≥ 15% compared to baseline levels)
Number of participants with complete TMA response status without the use of anti-C5 antibody therapy | Throughout the study duration, up to 4 years
  Complete thrombotic microangiopathy (TMA) Response is defined as (1) hematological normalization in platelet count (platelet count ≥150 x 109/L) and LDH (below ULN), and (2) improvement in kidney function (≥ 25% serum creatinine reduction from baseline or ≥ 25% serum creatinine reduction compared to serum creatinine values prior to initiation of anti-C5 antibody therapy)
Estimated glomerular filtration rate (eGFR) | Throughout study duration, up to 4 years
  Estimated glomerular filtration rate (eGFR) based on eGFR categories will be collected.
  Serum creatinine as measured in mg/dL as part of the clinical chemistry panel through the central laboratory will be used to calculate the eGFR applying the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
Chronic kidney disease (CKD) stage | Throughout study duration, up to 4 years
  Chronic kidney disease (CKD) stage (1-5) based on eGFR categories will be provided:
  * Stage 1 (G1): Kidney damage with normal kidney function
  * Stage 2 (G2): Mild loss of kidney function
  * Stage 3 (G3): 3a: Mild to moderate loss of kidney function; 3b: Moderate to severe loss of kidney function
  * Stage 4 (G4): Severe loss of kidney function
  * Stage 5 End stage renal disease (kidney failure): Kidney failure and need for transplant or dialysis
Number of participants by dialysis requirement status | Throughout the study duration, up to 4 years
  Dialysis requirement status will be provided
Number of participants with Thrombotic Microangiopathy (TMA) related adverse events | Throughout study duration, up to 4 years
  TMA related events during the study defined as any of the following:
  * Irreversible (>3 months) reduction in eGFR rate by ≥20%, not attributable to another cause
  * An episode of acute kidney injury (AKI) attributed to a TMA that requires renal replacement therapy
  * A non-renal manifestation of a TMA that requires hospitalization, or causes irreversible organ damage or death.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Brazil (2):
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Novartis Investigative Site, Beijing, China
- Novartis Investigative Site, Ostrava, Poruba, Czechia
- India (2):
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com